CLINICAL TRIAL: NCT01975298
Title: A Multinational, Multicenter, Randomized, Double-Blind, Parallel-Group, Active-Control (Rater Blinded) Study, to Evaluate The Efficacy, Safety And Tolerability Of 2 Doses Of Oral Administration Of Laquinimod (0.6 mg/Day Or 1.2 mg/Day) Compared to Interferon ß-1a Administered Intra Muscular Once Weekly in Subjects With Relapsing Remitting Multiple Sclerosis (RRMS).
Brief Title: A Study to Evaluate 2 Doses Of Oral Administration Of Laquinimod Compared to Interferon ß-1a Administered by Injection in Participants With Relapsing Remitting Multiple Sclerosis (RRMS)
Acronym: LIBRETTO
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAQ-MS-306; 2013-002082-19 (EudraCT Number)
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — laquinimod; Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Laquinimod 0.6 mg (Experimental)
  Interventions: Drug: Laquinimod
- Laquinimod 1.2 mg (Experimental)
  Interventions: Drug: Laquinimod
- Avonex® (Active Comparator)
  Interventions: Drug: Avonex®

INTERVENTIONS:
Drug: Laquinimod — Oral Administration
  Other Names: TV-5600
  Arms: Laquinimod 0.6 mg; Laquinimod 1.2 mg
Drug: Avonex® — Interferon β1A 30 μg/0.5mL administered Intra Muscular
  Other Names: Interferon β1A
  Arms: Avonex®

SUMMARY:
The purpose of the study is to assess the efficacy, safety, and tolerability of two doses of laquinimod compared to Avonex®

ELIGIBILITY:
Inclusion Criteria

* Subjects must have a confirmed and documented RRMS diagnosis as defined by the Revised McDonald criteria, with relapse onset disease or a relapsing-remitting disease course.
* Subjects must be ambulatory with an Kurtzke EDSS score of 0-5.5 at both Screening and Baseline (randomization) visits.
* Subjects must be in a stable neurological condition, relapse-free and free of any corticosteroid treatment (intravenous [IV], IM and/or per os [PO]) or adrenocorticotrophic hormone (ACTH), 60 days prior to randomization.
* Subjects must have experienced at least 1 documented relapse in the last year prior to randomization or 2 relapses in the last 3 years prior to randomization.
* Subjects must be between 18 and 55 years of age at screening, inclusive.
* Women of child-bearing potential must practice an acceptable method of birth control until 30 days after the last dose of treatment was administered (acceptable methods of birth control in this study include: surgical sterilization, intrauterine devices, oral contraceptive, contraceptive patch, long-acting injectable contraceptive or double-barrier method [condom or diaphragm with spermicide]).
* Subjects must be able to sign and date a written informed consent prior to entering the study.
* Subjects must be willing and able to comply with the protocol requirements for the duration of the study.

  * other criteria may apply, please contact the investigator for more information

Exclusion Criteria:

* Subjects with progressive forms of MS.
* Subjects with Neuromyelitis Optica (NMO).
* Use of experimental or investigational drugs and/or participation in drug clinical studies within 6 months prior to Baseline visit (randomization).
* Use of immunosuppressive agents, or cytotoxic agents, including cyclophosphamide and azatioprine within 12 months prior to Baseline.
* Natalizumab (Tysabri®) if given more than 6 months prior to randomization AND the subject is John Cunningham (JC) virus antibody test negative at Screening.
* Previous use of Rituximab, ocrelizumab, or ofatumumab is allowed if the B cell count (CD19) is higher than 80 cells /μL.
* Previous treatment with glatiramer acetate (Copaxone®e), fingolimod (Gilenya®), BG-12 (Tecfidera), Teriflunomide (Aubagio®) or intravenous immunoglobulin (IVIG) within 2 months prior to Baseline.
* Use of mitoxantrone (Novantrone) within 5 years prior to Screening. Use of mitoxantrone (Novantrone) >5 years before screening is allowed in subjects with normal ejection fraction and who did not exceed the total lifetime maximal dose.
* Chronic (more than 30 consecutive days or monthly dosing, eg, with the intent of MS disease modification) systemic (IV, IM or PO) corticosteroid treatment within 2 months prior to Baseline.
* Previous use of cladribine.
* Previous use of laquinimod or Avonex® IM.
* Treatment with other Interferon-β (either 1a subcutaneous [SC] or 1b SC) within 60 days before baseline (earlier treatment will be allowed if the reason for discontinuation was not treatment failure or for Interferon-β related safety reasons. This decision will be taken by the investigator).
* Previous total body irradiation or total lymphoid irradiation.
* Previous stem cell treatment, autologous bone marrow transplantation, or allogenic bone marrow transplantation.
* Acute infection within 2 weeks prior to Baseline visit.
* Major trauma or surgery within 2 weeks prior to Baseline visit.
* Use of moderate/strong inhibitors of CYP3A4 within 2 weeks prior to Baseline.
* Use of inducers of CYP3A4 within 2 weeks prior to Baseline
* Pregnancy or breast feeding.
* Serum levels ≥ 3 times (x) upper limit of normal (ULN) of either ALT or AST at Screening.
* Serum direct bilirubin ≥ 2xULN at Screening.
* Subjects with a clinically significant or unstable medical or surgical condition or any other condition that cannot be well-controlled by the allowed medications permitted in the study protocol that would preclude safe and complete study participation, as determined by medical history, physical examinations, ECG, laboratory tests MRI or chest X-ray
* Any acute pulmonary disorder.
* A central nervous system disorder other than MS that may jeopardize the participation in the study, including such disorders that are demonstrated on the baseline MRI.
* A gastrointestinal disorder that may affect the absorption of study medication.
* Renal disease.
* Thyroid disease: hyperthyroidism, hypothyroidism.
* Any form of acute or chronic liver disease.
* Known human immunodeficiency virus positive status.
* A clinical history of drug and/or alcohol abuse.
* Unstable psychiatric disorder.
* A history of seizure disorder, with the last convulsive episode within 12 months prior to Screening visit.
* Any malignancies, excluding basal cell carcinoma, in the 5 years prior to randomization.
* Twenty or more gadolinium - enhancing lesions on baseline MRI.
* A known history of sensitivity to gadolinium (Gd).
* GFR ≤ 60 mL/min at the screening visit.
* Inability to successfully/safely undergo MRI scanning.
* Subjects who underwent endovascular treatment for Chronic Cerebrospinal Venous Insufficiency (CCSVI).
* Known hypersensitivity that would preclude administration of laquinimod capsule, such as hypersensitivity to: mannitol, meglumine, or sodium stearyl fumarate.
* A known history of hypersensitivity to natural or recombinant interferon β, human albumin, or any other component of the formulation of Avonex®
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals

  * other criteria may apply, please contact the investigator for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Brain Atrophyas observed by Magnetic Resonance Imaging (MRI) | Baseline and Month 12.
  This is assessed by an MRI and is a measure of brain volume

SECONDARY OUTCOMES:
The cumulative number of reported influenza-like symptoms | Baseline to Month 3
Cumulative number of new T2 lesions observed by Magnetic Resonance Imaging (MRI) between the 2 laquinimod doses | Baseline, Month 6 and Month 12
Summary of Participant with Adverse Events | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.